CLINICAL TRIAL: NCT04588454
Title: 18F-PSMA PET/CT for Visualization of Glioblastoma Multiforme
Acronym: PSMA-GBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL64616.091.18
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-10

CONDITIONS: Glioblastoma Multiforme
Keywords: nuclear imaging; prostate specific membrane antigen; glioblastoma multiforme; positron emission tomography
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-PSMA-1007 PET/CT (Experimental)
  Interventions: Other: 18F-PSMA-1007 PET tracer

INTERVENTIONS:
Other: 18F-PSMA-1007 PET tracer — 18F-PSMA-1007 PET/CT

SUMMARY:
This is a pilot study to determine uptake of PET tracer 18F-PSMA-1007 in primary glioblastoma.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) is a highly vascularised tumour. Previous studies have shown that prostate-specific membrane antigen (PSMA) is robustly expressed by the tumour vascular endothelium of GBM and thus could be an interesting target for diagnosis and treatment.

Several groups have focused on the development of 18F-labeled PSMA ligands for PET imaging. 18F as a radionuclide has several advantages over 68Ga. Due to the longer half-life compared (110 min for 18F compared to 68 min for 68Ga) allows for centralized production and distribution to greater areas. Furthermore, multiple doses of 18F can be produced in one synthesis, while each gallium generator provides only one or two elutions per day. Moreover, due to the decreased positron energy (0.65 MeV for 18F compared to 1.90 MeV for 68Ga) imaging resolution may be higher. The first generation of 18F-PSMA ligands, such as 18F-DCFBC, suffered from high background due to slow blood clearance. The second generation 18F-DCFPyL PSMA ligand has a fast elimination via the urinary route and showed high tumor-to-blood ratios. Benesova et al developed the 177Lu-DKFZ-61, which is suitable for labelling with both diagnostic 68Ga as well as therapeutic 177Lu (beta-emitting) or 225Ac (alpha-emitting), and Giesel at al developed 18F-PSMA-1007, which is structurally related to DKZF-617.

Since various studies have shown feasibility of PSMA imaging in brain lesions of patients with recurrent GBM, we want to extend these results in a cohort of patients with a first-diagnosed suspected GBM. We want to use the PET tracer 18F-PSMA-1007. If this technique can be implemented successfully, the added value of 18F-PSMA PET/CT for tumour grading and differential diagnosis could be investigated further in larger patient cohorts (especially with recurrent brain lesions). These studies will pave the way for further studies involving 177Lu-PSMA-based therapy, which is currently applied in patients with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Suspected GBM on MRI scan
* Scheduled for tumor resection at Radboudumc
* Age ≥18 years

Exclusion Criteria:

* Age < 18 years
* Pregnancy or the wish to become pregnant within 6 months
* Creatinine clearance below 40ml/min
* Liver disease defined as aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
The uptake of 18F-PSMA PET/CT in suspected GBM lesions | uptake of the tracer at 2 hours post injection

SECONDARY OUTCOMES:
The correlation between PSMA protein and RNA expression with 18F-PSMA PET/CT uptake | uptake of the tracer at 2 hours post injection vs RNA expression determined from excised tumor tissue
Correlation between 18F-PSMA PET/CT and T1Gd MRI | Uptake of the tracer at 2 hours post injection vs pre-op MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McBriar JD, Shafiian N, Scharf S, Boockvar JA, Wernicke AG. Prostate-Specific Membrane Antigen Use in Glioma Management: Past, Present, and Future. Clin Nucl Med. 2024 Sep 1;49(9):806-816. doi: 10.1097/RLU.0000000000005365. Epub 2024 Jul 1. PMID 38968568